CLINICAL TRIAL: NCT02421744
Title: A Task-oriented Circuit Training in Multiple Sclerosis: a Multicentric Randomized Controlled Trial
Brief Title: A Task-oriented Circuit Training in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Studio multicentrico TOCT SM
Record Dates: First submitted 2015-01-19; First posted 2015-04-21 (Estimated); Last update posted 2018-11-29 (Actual); Status verified 2017-05

CONDITIONS: Multiple Sclerosis
Keywords: rehabilitation; Multiple Sclerosis; mobility; gait; task-oriented training
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Task Oriented Circuit Training (Experimental): TOCT includes six different workstations in which subjects exercise for 5 minutes in each one (3 minutes of exercise and 2 minutes of rest). During each session, subjects undergo 2 laps that take about 60 minutes (6 workstation × 5 minutes × 2 laps), with 10 minutes of rest after each lap. In addition, walking endurance is trained by 30 minutes walking on the treadmill including rests if necessary. This is a progressive circuit and subjects while exercising receive feedbacks (visual and auditory) by the physiotherapist. Rests are used to discuss about difficulties and to provide further feedbacks. One session includes up to 3 patients and lasts 120 minutes, 5 days/week for 2 weeks. After this period they will receive a home-exercise maintenance program for 3 months.
  Interventions: Behavioral: Task Oriented Circuit Training
- Delayed Onset TOCT (Active Comparator): The control group will not receive any specific rehabilitation treatment for gait performance and mobility improvement. At any case, the control group will be authorized, at will, to exercise in non-rehabilitative contexts (i.e. swimming, walking, yoga) for 14 weeks. After this period they will receive TOCT as treatment plus a home-exercise maintenance program for 3 months.
  Interventions: Behavioral: Delayed Onset TOCT

INTERVENTIONS:
Behavioral: Task Oriented Circuit Training — TOCT includes six different workstations in which subjects exercise for 5 minutes in each one (3 minutes of exercise and 2 minutes of rest). During each session, subjects undergo 2 laps that take about 60 minutes (6 workstation × 5 minutes × 2 laps), with 10 minutes of rest after each lap. In addition, walking endurance is trained by 30 minutes walking on the treadmill including rests if necessary. This is a progressive circuit and subjects while exercising receive feedbacks (visual and auditory) by the physiotherapist. Rests are used to discuss about difficulties and to provide further feedbacks. One session includes up to 3 patients and lasts 120 minutes, 5 days/week for 2 weeks. After this period they will receive a home-exercise maintenance program for 3 months.
  Arms: Task Oriented Circuit Training
Behavioral: Delayed Onset TOCT — The control group will not receive any specific rehabilitation treatment for gait performance and mobility improvement. At any case, the control group will be authorized, at will, to exercise in non-rehabilitative contexts (i.e. swimming, walking, yoga) for 14 weeks. After this period they will receive TOCT as treatment plus a home-exercise maintenance program for 3 months.
  Arms: Delayed Onset TOCT

SUMMARY:
Our primary hypothesis is that a two weeks high-intensity task-oriented circuit training followed by a structured 3 months home exercise program would have higher benefits compared to a delayed-treatment group as control in people with multiple sclerosis and mild to moderate gait impairment.

Our secondary hypothesis is that there could be retention of clinical gains in subjects that underwent TOCT plus structured 3 months home exercise program.

DETAILED DESCRIPTION:
This is a single blind randomized-controlled trial to test the effects of a task oriented training on locomotor function, mobility and balance in multiple sclerosis subjects with mild to moderate gait impairments (EDSS 4-5.5).

Subjects and methods:54 multiple sclerosis patients will be recruited in two outpatient rehabilitation clinics (Azienda Ospedaliero- Universitaria di Ferrara and Azienda Ospedaliero-Universitaria Pisana). Informed consent will be obtained. Participants enrolled will be included in 2 different treatment groups: experimental group will receive 10 TOCT sessions over 2 weeks (2 hours/each session) followed by a 3 months home exercise program, whereas control group will be included into a delayed-treatment group. Three subjects with a supervisor physiotherapist will take part at the TOCT. Primary outcome measure will be walking endurance (Six Minute Walking Test); as secondary outcome we will test gait speed (Timed 25-Foot Walk), balance (Dynamic Gait Index) and mobility (Time Up and Go Test); through self-assessment questionnaires we will evaluate motor fatigue (Modified Fatigue Impact Scale - MFIS), walking ability (Multiple Sclerosis Walking Scale - 12), health-related quality of life (Multiple Sclerosis Impact Scale - 29 and Functional Assessment of Multiple Sclerosis). In addition to clinical outcomes, in a convenience sample we will have: (i) balance assessment (force platform); (ii) motorcortex oxygenation during walking (fNIRS); (iii) muscle oxygenation (NIRS); (iv) force and EMG signal; (v) mechanical and electrical fatigue assessment; (vi) brain connectivity (EEG). Outcome measures will be assessed 1 week prior to treatment initiation (T0), after two weeks to treatment initiation (T1), after the 3 months exercise program (T2) and at 3 months follow-up (T3) to evaluate treatments retention, by a clinician blinded to the treatment.

The specific aims will be (i) to test the effects on walking, mobility, balance, fatigue and health-related quality of life; (ii) to test the effects on cerebral oxygenation (fNIRS) during walking; (iii) muscle oxygenation (NIRS); (iv) force and EMG signal; (v) Mechanical and electrical fatigue assessment; (vi) brain connectivity (EEG) and (vii) to investigate the 3 months home exercise program's feasibility, satisfaction and adherence.

ELIGIBILITY:
Inclusion Criteria:

* males and females,
* community dwelling,
* age >18 and <75
* diagnosis of multiple sclerosis in a stable phase, with relapses > 3 months prior to study enrollment
* moderate gait impairments referred to Expanded Disability Status Scale (EDSS) between 4 and 5,5
* MMSE >24

Exclusion Criteria:

* neurologic conditions in addition to multiple sclerosis that may affect motor function
* medical conditions likely to interfere with the ability to safely complete the study
* pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-03; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Six-Minute Walking Test | Weeks: 0,2,14, 26
  The walking endurance is measured with the Six-Minute Walking Test. Subjects are instructed to walk up and down as far as possible a 22m walkway in six minutes, with the possibility to slow down and rest if necessary.

SECONDARY OUTCOMES:
Timed 25-Foot walk (25FWT) | weeks: 0,2,14, 26
  a quantitative measure of lower extremity function, also included in the Multiple Sclerosis Functional Composite (MSFC) . The patient is directed to one end of a clearly marked 25-foot course and is instructed to walk 25 feet (7.62m) as quickly as possible, but safely, using the prescribed assistive devices. The task is immediately administered again by having the patient walk back the same distance. Test will be performed according to the instructions reported on the manual of the National Multiple Sclerosis Society .
Time Up and Go Test | weeks: 0,2,14, 26
  Subjects will be given verbal instruction to stand up from a chair, walk 3 meters, cross a line marked on the floor, turn around, walk back, and sit down. A study staff member will guard the subject during the test. Subjects will perform 3 trials and the time it takes to perform each trial will be recorded with a stopwatch.
Dynamic Gait Index (DGI) | weeks: 0,2,14, 26
  Assesses individual's ability to modify balance while walking in the presence of external demands
Modified fatigue impact scale (MFIS) | weeks: 0,2,14, 26
  The MFIS is a modified form of the Fatigue Impact Scale (Fisk et al, 1994) based on items derived from interviews with MS patients concerning how fatigue impacts their lives. This instrument provides an assessment of the effects of fatigue in terms of physical, cognitive, and psychosocial functioning.
Multiple Sclerosis Walking Scale - 12 (MSWS-12) | weeks: 0,2,14, 26
  The 12-item multiple sclerosis walking scale (MSWS-12) is a self-report measure of the impact of MS on the individual's walking ability.
Multiple Sclerosis Impact Scale- 29 (MSIS-29) | weeks: 0,2,14, 26
  This is an health-rated quality of life questionnaire that assesses the impact of MS on physical and psychological functions. It is formed by 29 items on ADL I and II: 20 about physical activity and 9 of psychological status of the person. Each item can be scored with a value from 0 to 5; total score is given by the sum of all the items and then is transformed in a range from 0 to 100. A higher value correspond to a worse perception of subject's HRQoL.
Functional Assessment of Multiple Sclerosis (FAMS) | weeks: 0,2,14, 26
  Quality of life instrument of for use in people with MS. Consists of 59 items (44 of which are scored) in six quality of life domains. Higher scores indicate better quality of life.
Metabolic cerebral measurements by Near infrared spectroscopy | weeks: 0,2,14, 26
  Near InfraRed Spectroscopy (NIRS) is a noninvasive, portable technique for ambulatory or remote monitoring of human motor-cortex oxygenation changes in response to motor tasks. Patients will walk on the treadmill at a speed of 0.2 km/h assisted by personnel and with partial body weight support, performing 4 short tasks (30 seconds of walking) alternated by rest periods (30 seconds).
Postural sway (Center of pressure (COP) trajectories) | weeks: 0,2,14, 26
  Center of pressure (COP) trajectories
Force and EMG signal (perform an isometric extension of the knees on an isokinetic dynamometer (PrimusRS BTETM Technology), achieving their own Maximum Voluntary Contraction (MVC) | weeks: 0,2,14, 26
  Patients will perform an isometric extension of the knees on an isokinetic dynamometer (PrimusRS BTETM Technology), achieving their own Maximum Voluntary Contraction (MVC) during a set of 3 seconds trials.
Mechanical and electrical fatigue assessment (evaluated measuring sustained contractions in isometric tasks in lower limbs on an isokinetic dynamometer (PrimusRS BTETM Technology) | weeks: 0,2,14, 26
  Muscle fatigue will be evaluated measuring sustained contractions in isometric tasks in lower limbs on an isokinetic dynamometer (PrimusRS BTETM Technology), maintaining a MVC for knee and ankle extension for 60 s.
Brain plasticity and connectivity (High density EEG and vertical electrooculogram (EOG) will be recorded with a standard bipolar 64-channels montage and a DC-coupled amplifier (Micromed SD MRI, System Plus acquisition software) | weeks: 0,2,14, 26
  High density EEG and vertical electrooculogram (EOG) will be recorded with a standard bipolar 64-channels montage and a DC-coupled amplifier (Micromed SD MRI, System Plus acquisition software).
Metabolic muscular measurements by Near infrared spectroscopy | weeks: 0,2,14, 26
  Noninvasive muscle measurements will be performed at gastrocnemius by an optical imaging system consisting of 2 light source fibers and 2 detector fibers.

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Straudi, MD, Principal Investigator — Ferrara Rehabilitation Hospital
Locations (2):
- Italy (2):
  - Ferrara University Hospital, Ferrara
  - Azienda Ospedaliera Universitaria Pisana, Pisa